CLINICAL TRIAL: NCT04611295
Title: TELENeurological Evaluation and Support for the Emergency Department (TELENS-ED): an Open-label Clinical Trial
Brief Title: TELENeurological Support for Emergency Department
Acronym: TELENS-ED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Collaborators: Azienda USL Modena (Other)
Responsible Party: Principal Investigator, Stefano Meletti, Study coordinator and Clinical Investigator, Azienda Ospedaliero-Universitaria di Modena
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 942/2020/DISP/AOUMO
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Emergencies; Neurologic Disorder
MeSH Terms: conditions — Emergencies; Nervous System Diseases | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teleneurological evaluation and support (Experimental): teleneurological evaluation using a medical device certified as telemedicine system
  Interventions: Procedure: Teleneurological evaluation and support

INTERVENTIONS:
Procedure: Teleneurological evaluation and support — The study is aimed at developing a remote neurological consultancy system (teleconsultation) for patients with acute neurological symptoms in charge of hospital facilities without 24-hour availability of neurologist consultant.

SUMMARY:
Open-label, non-inferiority, teleconsultation with televisit study to compare efficacy, safety and users satisfaction of a TeleNeurological Support versus "in person" neurological examination in the emergency department

DETAILED DESCRIPTION:
The investigtors are going to perform an interventional, open-label study on the use of teleconsultation in the emergency department focused on neurological diseases other than stroke (for which a specific protocol already exists) in two Hospitals of Modena province, Italy.

The study is aimed at developing a remote neurological consultancy system (teleconsultation) for patients with acute neurological symptoms in charge of hospital facilities without 24-hour availability of neurologist consultant.

Pilot project setting: a) ED of Modena Policlinico Hospital in the afternoon, night, and public holidays, time windows in which the Neurologist consultant is not present at Policlinico Hospital; b) ED of Mirandola Hospital.

The project (enrolment) is expected to be developed over a period of 6 months in which 100 patients will be enrolled.

The primary objective is to assess whether a TeleNeurological Evaluation and Support for the Emergency Department can guarantee a faster but qualitatively not inferior diagnostic/therapeutic work-up if compared with in person examination, assuring the availability of all the necessary examinations and treatments with a consistent time reduction.

Secondary objectives: to determine if the usage of a teleconsultation physician for neurological evaluation compared to a conventional physician "de visu" in urgent but non-life-threatening neurological cases, is superior regarding 1) effect evaluation, 2) process evaluation, and 3) cost-benefit analysis.

Outcome and process indicators will be assessed and compared in the following groups:

* Experimental group (cases): a) patients who access the Policlinico Hospital ED in the afternoon and night-time and on holidays; b) patients who access the Mirandola Hospital ED during the period of the study.
* Control Groups: a) retrospectively collected data on neurological consultation performed by OCB Neurology for Policlinico Hospital patients in the same time slots in the same months of the last two years.; b) retrospectively collected data on neurological consultation performed by Carpi Neurology for Mirandola Hospital patients in the same time slots in the same months of the last two years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years
* Symptoms related to possible acute / subacute neurological pathology, or worsening of known neurological pathology, for which the ED physician considers neurological consultation indicated / necessary.
* Signing of informed consent to remote neurological evaluation.

Exclusion Criteria:

* All life-threatening emergency cases, where the study procedure would interfere with clinical practice
* Patients with known neurological pathology or with clinical severity to such an extent that the need for admission to OCB/Carpi Neurology unit or to the internal wards of the Policlinico is immediately evident.
* Refusal of the patient/caregiver to perform remote neurological evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Teleconsultation clinical application | 6 months
  Percentage of patients who undergo neurological teleconsultation over the number of patients who access on the days and in the time slots in which the service is active and needing a neurological evaluation.
Teleconsultation diagnostic efficacy | 6 months
  Percentage of patients re-admitted to the ED in the 7 days following the date of neurological consultation. It is expected that for the patients of the neurological teleconsultation the % of re-admission to ED will not exceed that of the patients undergone standard neurological advice.
Teleconsultation efficacy - hospitalization | 6 months
  Percentage of hospitalized patients among those undergone TeleNeurology compared to percentage of hospitalization for patients with in person neurological evaluation. It is expected that for patients of the teleneurology group the % of hospitalization will not exceed that of patients undergone standard neurological advice.
Time 'door to end of diagnostic process' | 6 months
  The total time from ED admission to the end of the diagnostic and therapeutic process (time spent in the ED): this time is expected to be significantly shorter for patients in the teleneurology group than for patients having a standard neurological advice.
Time 'door to end of neurological evaluation' | 6 months
  The time from the ED admission to the end of the remote neurological consultation: this time is expected to be significantly shorter for patients in the teleneurology group than for patients having a standard neurological advice

SECONDARY OUTCOMES:
Cost-effectiveness | 6 months
  Evaluation of costs, or cost-effectiveness. For the evaluation of costs, it will be developed a model that considers the cost of the system on the one hand, and the savings in terms of personnel (medical personnel, paramedics and ambulances costs). Outcome indicator.
Evaluation of the level of satisfaction of the users | 6 months
  For this purpose an evaluation form will be provided to patients / family members. Users satisfaction will be measured by visual analogue scale (VAS) where 100 is the highest satisfaction and 0 is the lowest. Outcome indicator.
Evaluation of the level of satisfaction of the health personnel. | 6 months
  For this purpose an evaluation form will be provided to medical personnel involved. Personnel satisfaction will be measured by visual analogue scale (VAS) where 100 is the highest satisfaction and 0 is the lowest. Outcome indicator.
Teleconsultation failure | 6 months
  Percentage of cases assessed by teleconsultation for which the neurologist was unable to make remote decisions and requested for sending the patient to Hub Hospital for a "first-person" evaluation. Process indicator.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Luciani, MD, Principal Investigator — Azienda Ospedaliero Universitaria Policlinico Modena
Locations (2):
- Italy (2):
  - Azienda USL di Modena, Modena
  - Azienda Ospedaliero Universitaria di Modena, Modena

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available at study end
Access Criteria: Upon request to principal investigator

REFERENCES:
- [Background] Piano per il miglioramento dell'accesso in Emergenza Urgenza nelle strutture sanitarie dell'Emilia-Romagna; https://bur.regione.emilia-romagna.it/dettaglio-inserzione?i=7b644492dfe2471787f041d37a19f2e8; 24.07.2019
- [Background] WHO. A health telematics policy in support of WHO's Health-For-All strategy for global health development: report of the WHO group consultation on health telematics, 11-16 December, Geneva, 1997. Geneva, World Health Organization, 1998.).
- [Background] Bove AA, Homko CJ, Santamore WP, Kashem M, Kerper M, Elliott DJ. Managing hypertension in urban underserved subjects using telemedicine--a clinical trial. Am Heart J. 2013 Apr;165(4):615-21. doi: 10.1016/j.ahj.2013.01.004. Epub 2013 Mar 6. PMID 23537980
- [Background] Verhoeven F, van Gemert-Pijnen L, Dijkstra K, Nijland N, Seydel E, Steehouder M. The contribution of teleconsultation and videoconferencing to diabetes care: a systematic literature review. J Med Internet Res. 2007 Dec 14;9(5):e37. doi: 10.2196/jmir.9.5.e37. PMID 18093904
- [Background] Brebner JA, Brebner EM, Ruddick-Bracken H. Accident and emergency teleconsultation for primary care--a systematic review of technical feasibility, clinical effectiveness, cost effectiveness and level of local management. J Telemed Telecare. 2006;12 Suppl 1:5-8. doi: 10.1258/135763306777978542. PMID 16884562
- [Background] Hersh W, Helfand M, Wallace J, Kraemer D, Patterson P, Shapiro S, Greenlick M. A systematic review of the efficacy of telemedicine for making diagnostic and management decisions. J Telemed Telecare. 2002;8(4):197-209. doi: 10.1258/135763302320272167. PMID 12217102
- [Background] Hersh WR, Hickam DH, Severance SM, Dana TL, Pyle Krages K, Helfand M. Diagnosis, access and outcomes: Update of a systematic review of telemedicine services. J Telemed Telecare. 2006;12 Suppl 2:S3-31. doi: 10.1258/135763306778393117. PMID 16989671
- [Background] Deldar K, Bahaadinbeigy K, Tara SM. Teleconsultation and Clinical Decision Making: a Systematic Review. Acta Inform Med. 2016 Jul 16;24(4):286-292. doi: 10.5455/aim.2016.24.286-292. PMID 27708494
- [Background] Nerlich M, Balas EA, Schall T, Stieglitz SP, Filzmaier R, Asbach P, Dierks C, Lacroix A, Watanabe M, Sanders JH, Doarn CR, Merrell RC; G8 Global Health Applications Subproject 4. Teleconsultation practice guidelines: report from G8 Global Health Applications Subproject 4. Telemed J E Health. 2002 Winter;8(4):411-8. doi: 10.1089/15305620260507549. PMID 12626110
- [Background] Epstein RM. Communication between primary care physicians and consultants. Arch Fam Med. 1995 May;4(5):403-9. doi: 10.1001/archfami.4.5.403. PMID 7742962
- [Background] Belyansky I, Martin TR, Prabhu AS, Tsirline VB, Howley LD, Phillips R, Sindram D, Heniford BT, Stefanidis D. Poor resident-attending intraoperative communication may compromise patient safety. J Surg Res. 2011 Dec;171(2):386-94. doi: 10.1016/j.jss.2011.04.011. Epub 2011 May 6. PMID 21601875
- [Background] Audebert HJ, Kukla C, Clarmann von Claranau S, Kuhn J, Vatankhah B, Schenkel J, Ickenstein GW, Haberl RL, Horn M; TEMPiS Group. Telemedicine for safe and extended use of thrombolysis in stroke: the Telemedic Pilot Project for Integrative Stroke Care (TEMPiS) in Bavaria. Stroke. 2005 Feb;36(2):287-91. doi: 10.1161/01.STR.0000153015.57892.66. Epub 2004 Dec 29. PMID 15625294
- [Background] Audebert HJ, Schenkel J, Heuschmann PU, Bogdahn U, Haberl RL; Telemedic Pilot Project for Integrative Stroke Care Group. Effects of the implementation of a telemedical stroke network: the Telemedic Pilot Project for Integrative Stroke Care (TEMPiS) in Bavaria, Germany. Lancet Neurol. 2006 Sep;5(9):742-8. doi: 10.1016/S1474-4422(06)70527-0. PMID 16914402
- [Background] Audebert HJ, Schultes K, Tietz V, Heuschmann PU, Bogdahn U, Haberl RL, Schenkel J; Telemedical Project for Integrative Stroke Care (TEMPiS). Long-term effects of specialized stroke care with telemedicine support in community hospitals on behalf of the Telemedical Project for Integrative Stroke Care (TEMPiS). Stroke. 2009 Mar;40(3):902-8. doi: 10.1161/STROKEAHA.108.529255. Epub 2008 Nov 20. PMID 19023095
- [Background] Demaerschalk BM, Bobrow BJ, Raman R, Kiernan TE, Aguilar MI, Ingall TJ, Dodick DW, Ward MP, Richemont PC, Brazdys K, Koch TC, Miley ML, Hoffman Snyder CR, Corday DA, Meyer BC; STRokE DOC AZ TIME Investigators. Stroke team remote evaluation using a digital observation camera in Arizona: the initial mayo clinic experience trial. Stroke. 2010 Jun;41(6):1251-8. doi: 10.1161/STROKEAHA.109.574509. Epub 2010 Apr 29. PMID 20431081
- [Background] Handschu R, Scibor M, Willaczek B, Nuckel M, Heckmann JG, Asshoff D, Belohlavek D, Erbguth F, Schwab S; STENO Project. Telemedicine in acute stroke: remote video-examination compared to simple telephone consultation. J Neurol. 2008 Nov;255(11):1792-7. doi: 10.1007/s00415-008-0066-9. Epub 2008 Dec 8. PMID 19156491
- [Background] Meyer BC, Raman R, Hemmen T, Obler R, Zivin JA, Rao R, Thomas RG, Lyden PD. Efficacy of site-independent telemedicine in the STRokE DOC trial: a randomised, blinded, prospective study. Lancet Neurol. 2008 Sep;7(9):787-95. doi: 10.1016/S1474-4422(08)70171-6. PMID 18676180
- [Background] Sejersten M, Sillesen M, Hansen PR, Nielsen SL, Nielsen H, Trautner S, Hampton D, Wagner GS, Clemmensen P. Effect on treatment delay of prehospital teletransmission of 12-lead electrocardiogram to a cardiologist for immediate triage and direct referral of patients with ST-segment elevation acute myocardial infarction to primary percutaneous coronary intervention. Am J Cardiol. 2008 Apr 1;101(7):941-6. doi: 10.1016/j.amjcard.2007.11.038. Epub 2008 Jan 25. PMID 18359312
- [Background] Chua R, Craig J, Wootton R, Patterson V. Randomised controlled trial of telemedicine for new neurological outpatient referrals. J Neurol Neurosurg Psychiatry. 2001 Jul;71(1):63-6. doi: 10.1136/jnnp.71.1.63. PMID 11413265
- [Background] Skorning M, Bergrath S, Rortgen D, Brokmann JC, Beckers SK, Protogerakis M, Brodziak T, Rossaint R. [E-health in emergency medicine - the research project Med-on-@ix]. Anaesthesist. 2009 Mar;58(3):285-92. doi: 10.1007/s00101-008-1502-z. German. PMID 19221700
- [Background] Ziegler V, Rashid A, Muller-Gorchs M, Kippnich U, Hiermann E, Kogerl C, Holtmann C, Siebler M, Griewing B. [Mobile computing systems in preclinical care of stroke. Results of the Stroke Angel initiative within the BMBF project PerCoMed]. Anaesthesist. 2008 Jul;57(7):677-85. doi: 10.1007/s00101-008-1395-x. German. PMID 18542893
- [Background] Tso JV, Farinpour R, Chui HC, Liu CY. A Multidisciplinary Model of Dementia Care in an Underserved Retirement Community, Made Possible by Telemedicine. Front Neurol. 2016 Dec 23;7:225. doi: 10.3389/fneur.2016.00225. eCollection 2016. PMID 28066313
- [Background] Rasmusson KA, Hartshorn JC. A comparison of epilepsy patients in a traditional ambulatory clinic and a telemedicine clinic. Epilepsia. 2005 May;46(5):767-70. doi: 10.1111/j.1528-1167.2005.44804.x. PMID 15857445
- [Background] Muller KI, Alstadhaug KB, Bekkelund SI. A randomized trial of telemedicine efficacy and safety for nonacute headaches. Neurology. 2017 Jul 11;89(2):153-162. doi: 10.1212/WNL.0000000000004085. Epub 2017 Jun 14. PMID 28615434
- [Background] Dorsey ER, Deuel LM, Voss TS, Finnigan K, George BP, Eason S, Miller D, Reminick JI, Appler A, Polanowicz J, Viti L, Smith S, Joseph A, Biglan KM. Increasing access to specialty care: a pilot, randomized controlled trial of telemedicine for Parkinson's disease. Mov Disord. 2010 Aug 15;25(11):1652-9. doi: 10.1002/mds.23145. PMID 20533449
- [Background] AAN Recommendations for Expanded Coverage of Telemedicine Services. Updated on 1st July, 2020. https://www.aan.com/siteassets/home-page/tools-and-resources/practicing-neurologist--administrators/practice-top-5/aan-comments-to-cms-telemed-coverage.pdf
- [Background] Cohen BH, Busis NA, Ciccarelli L. Coding in the World of COVID-19: Non-Face-to-Face Evaluation and Management Care. Continuum (Minneap Minn). 2020 Jun;26(3):785-798. doi: 10.1212/CON.0000000000000874. PMID 32487907
- [Background] George BP, Kelly AG. Rethinking Regional Neurologic Care in the Coronavirus Disease 2019 Era. JAMA Neurol. 2020 Sep 1;77(9):1061-1062. doi: 10.1001/jamaneurol.2020.1956. No abstract available. PMID 32597937
- [Background] von Oertzen TJ, Macerollo A, Leone MA, Beghi E, Crean M, Oztuk S, Bassetti C, Twardzik A, Bereczki D, Di Liberto G, Helbok R, Oreja-Guevara C, Pisani A, Sauerbier A, Sellner J, Soffietti R, Zedde M, Bianchi E, Bodini B, Cavallieri F, Campiglio L, Maia LF, Priori A, Rakusa M, Taba P, Moro E, Jenkins TM; EANcore COVID-19 task force. EAN consensus statement for management of patients with neurological diseases during the COVID-19 pandemic. Eur J Neurol. 2021 Jan;28(1):7-14. doi: 10.1111/ene.14521. Epub 2020 Oct 15. PMID 33058321
- [Background] Dorsey ER, Topol EJ. State of Telehealth. N Engl J Med. 2016 Jul 14;375(2):154-61. doi: 10.1056/NEJMra1601705. No abstract available. PMID 27410924
- [Background] Czeisler ME, Marynak K, Clarke KEN, Salah Z, Shakya I, Thierry JM, Ali N, McMillan H, Wiley JF, Weaver MD, Czeisler CA, Rajaratnam SMW, Howard ME. Delay or Avoidance of Medical Care Because of COVID-19-Related Concerns - United States, June 2020. MMWR Morb Mortal Wkly Rep. 2020 Sep 11;69(36):1250-1257. doi: 10.15585/mmwr.mm6936a4. PMID 32915166
- [Background] Lange SJ, Ritchey MD, Goodman AB, Dias T, Twentyman E, Fuld J, Schieve LA, Imperatore G, Benoit SR, Kite-Powell A, Stein Z, Peacock G, Dowling NF, Briss PA, Hacker K, Gundlapalli AV, Yang Q. Potential Indirect Effects of the COVID-19 Pandemic on Use of Emergency Departments for Acute Life-Threatening Conditions - United States, January-May 2020. MMWR Morb Mortal Wkly Rep. 2020 Jun 26;69(25):795-800. doi: 10.15585/mmwr.mm6925e2. PMID 32584802
- [Background] Teo KC, Leung WCY, Wong YK, Liu RKC, Chan AHY, Choi OMY, Kwok WM, Leung KK, Tse MY, Cheung RTF, Tsang AC, Lau KK. Delays in Stroke Onset to Hospital Arrival Time During COVID-19. Stroke. 2020 Jul;51(7):2228-2231. doi: 10.1161/STROKEAHA.120.030105. Epub 2020 May 20. PMID 32432998
- [Background] Keesara S, Jonas A, Schulman K. Covid-19 and Health Care's Digital Revolution. N Engl J Med. 2020 Jun 4;382(23):e82. doi: 10.1056/NEJMp2005835. Epub 2020 Apr 2. No abstract available. PMID 32240581
- [Derived] Mandrioli J, Santangelo M, Luciani A, Toscani S, Zucchi E, Giovannini G, Martinelli I, Cecoli S, Bigliardi G, Scanavini S, Meletti S. TeleNeurological evaluation and Support for the Emergency Department (TeleNS-ED): protocol for an open-label clinical trial. BMJ Open. 2021 May 19;11(5):e048293. doi: 10.1136/bmjopen-2020-048293. PMID 34011601